CLINICAL TRIAL: NCT04380766
Title: Effects of Covid-19 Pandemic on Pancreatic Surgery in Italy. A Multicenter Observational Clinical Study
Brief Title: Covid-19 Pandemic and Pancreatic Surgery in Italy
Acronym: PanCOVID
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Sergio Alfieri, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: FPGemelliIRCCS
Record Dates: First submitted 2020-04-21; First posted 2020-05-08 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Pancreatic surgery; COVID-19
MeSH Terms: conditions — Pancreatic Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-COVID: All patients with pancreatic cancer diagnosis before COVID-19 pandemic
  Interventions: Procedure: Evaluation of changes in the diagnostic-therapeutic pathway for patients affected by pancreatic cancer
- COVID: All patients with pancreatic cancer diagnosis during COVID-19 pandemic
  Interventions: Procedure: Evaluation of changes in the diagnostic-therapeutic pathway for patients affected by pancreatic cancer

INTERVENTIONS:
Procedure: Evaluation of changes in the diagnostic-therapeutic pathway for patients affected by pancreatic cancer — Comparison between the pre-COVID and COVID groups of general, clinical, endoscopic and surgical outcomes

SUMMARY:
Pancreatic cancer (PC) is recognized as one of the most challenging tumors to deal with and it is still characterized by a poor long-term prognosis. However, treatment of PC in high-volume centers with the support of a multidisciplinary approach has widely demonstrated improvement both in terms of short- and long-term outcomes. The recent worldwide spread of Covid-19 pandemic significantly affected the healthcare systems of most countries in the world, particularly in red areas such as Italy, with more than 100.000 cases in a two-month time lapse. This inevitably reflected in a reorganization of hospital activities, including the diagnostic and therapeutic pathways for PC treatment. With the aim of giving an objective and real representation of the impact of Covid-19 on PC treatment, the investigator here propose a multicenter Italian observational study comparing a 6-month period before and during the Covid-19 pandemic. Only high-volume centers will be involved in the study. A comparison between the general, clinical, endoscopic and surgical outcomes will be performed by means of a global and month-by-month analysis between the two study periods.

ELIGIBILITY:
Inclusion Criteria:

all patients with a diagnosis of pancreatic cancer referred to one of the centers involved in the study during the two study periods

Exclusion Criteria:

* patients under the age of 18
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with diagnosis of pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in pancreatic cancer management during the COVID-19 pandemic | From admission to discharge/last outpatient visit, whichever comes first, assessed up to the 30th of June 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS di Roma, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quero G, Pecorelli N, Paiella S, Fiorillo C, Petrone MC, Rosa F, Capretti G, Laterza V, Kauffmann E, Nobile S, Butturini G, Ferrari G, Coratti A, Casadei R, Mazzaferro V, Boggi U, Zerbi A, Salvia R, Falconi M, Alfieri S. Quantitative assessment of the impact of COVID-19 pandemic on pancreatic surgery: an Italian multicenter analysis of 1423 cases from 10 tertiary referral centers. Updates Surg. 2022 Feb;74(1):255-266. doi: 10.1007/s13304-021-01171-8. Epub 2021 Nov 24. PMID 34817837